CLINICAL TRIAL: NCT06981936
Title: Evaluation of Balance Tablets in Reducing Vitamin and Mineral Deficiencies in Patients Using GLP-1 Receptor Agonists for Weight Loss
Brief Title: This Randomized Trial Aims to Investigate the Efficacy of Balanced Nutritional Tablets-Comprehensive Multivitamin and Mineral Supplements- in Preventing Micronutrient Deficiencies Among Patients Utilizing GLP-1 RAs for Weight Loss in Comparison to a Placebo Control
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, Surgeon, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Balance tablets And GLP1
Record Dates: First submitted 2025-05-11; First posted 2025-05-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Micronutrient Deficiencies
Keywords: Balance Tablets; Vitamin and Mineral Deficiencies; GLP-1 Receptor Agonists for Weight Loss; Weight Loss; Micronutrient Deficiencies
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention arms:
  * Intervention (Balance Tablet) Group: Participants take one Balance multivitamin/mineral tablet daily for 12 months. Each Balance tablet contains a broad range of vitamins and trace minerals at doses designed to prevent deficiencies (including but not limited to vitamins A, B-complex, C, D, E, K, calcium, iron, zinc, magnesium, selenium, and others, per standard multivitamin composition).
  * Control (Placebo) Group: Participants take one placebo tablet daily for 12 months. The placebo is an inert pill formulated to be indistinguishable from the Balance tablet in appearance, weight, and taste.
  * All participants will continue their prescribed GLP-1 RA therapy and any standard dietary advice for weight loss as per their treating provider. Compliance will be encouraged through monthly reminders and pill count checks; participants will be asked to return unused tablets at each study visit to monitor adherence.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Balance Tablet) Group (Experimental): Participants take one Balance multivitamin/mineral tablet daily for 12 months. Each Balance tablet contains a broad range of vitamins and trace minerals at doses designed to prevent deficiencies (including but not limited to vitamins A, B-complex, C, D, E, K, calcium, iron, zinc, magnesium, selenium, and others, per standard multivitamin composition).
  Interventions: Drug: Balance Tablet
- Control (Placebo) Group (Placebo Comparator): Participants take one placebo tablet daily for 12 months. The placebo is an inert pill formulated to be indistinguishable from the Balance tablet in appearance, weight, and taste.
  Interventions: Drug: Control (placebo)

INTERVENTIONS:
Drug: Balance Tablet — Each Balance tablet contains a broad range of vitamins and trace minerals at doses designed to prevent deficiencies (including but not limited to vitamins A, B-complex, C, D, E, K, calcium, iron, zinc, magnesium, selenium, and others, per standard multivitamin composition).
  Arms: Intervention (Balance Tablet) Group
Drug: Control (placebo) — The placebo is an inert pill formulated to be indistinguishable from the Balance tablet in appearance, weight, and taste.
  Arms: Control (Placebo) Group

SUMMARY:
Glucagon-like peptide-1 receptor agonists (GLP-1 RAs), including Ozempic (semaglutide) and Saxenda (liraglutide), are gaining traction in treating obesity and its associated diseases due to their capacity to facilitate substantial weight loss through mechanisms such as appetite suppression and delayed gastric emptying. Clinical trials have consistently shown that patients prescribed GLP-1 RAs can achieve significant body weight reductions when combined with appropriate dosing and lifestyle modifications.

However, the chronic appetite suppression and reduced caloric intake associated with prolonged GLP-1 RA use may increase the risk of micronutrient deficiencies, paralleling the biochemical changes observed after metabolic and bariatric surgery (MBS). In MBS cohorts, insufficient dietary intake coupled with malabsorption frequently results in deficiencies of essential vitamins and minerals, even in patients adhering to standard multivitamin regimens.

Research has demonstrated that high-dose specialized multivitamin supplementation can substantially lower the incidence of postoperative micronutrient deficiencies in MBS patients. This raises the possibility that proactive nutrient supplementation might similarly benefit individuals undergoing weight loss with GLP-1 RAs, although this hypothesis remains to be empirically validated.

To address this gap, this randomized trial aims to investigate the efficacy of Balanced nutritional tablets-comprehensive multivitamin and mineral supplements- in preventing micronutrient deficiencies among patients utilizing GLP-1 RAs for weight loss in comparison to a placebo control. Moreover, the study will assess changes in key nutrient biomarkers and relevant clinical outcomes over 12 months.

DETAILED DESCRIPTION:
Primary Objectives:

• Evaluate the efficacy of daily Balance multivitamin tablets in reducing the incidence of vitamin and mineral deficiencies among patients undergoing treatment with GLP-1 receptor agonists (RAs) for weight loss over 12 months, in comparison to a placebo group.

Secondary Objectives:

* Assessment of changes in serum concentrations of key vitamins and minerals such as vitamin B12, 25-hydroxyvitamin D, ferritin, and folate.
* comparing data collected at baseline with that gathered at the 12-month mark between the Balance multivitamin and placebo groups.
* Evaluate the effects of the intervention on body weight and various anthropometric measures, including Body Mass Index (BMI), percent excess weight loss (%EWL), and percent total body weight loss (%TWL), over the same 12-month period.
* Investigate the occurrence of hypervitaminosis, defined as elevated vitamin levels above normal ranges, within both intervention groups.
* Monitor adherence to the daily tablet regimen, ensuring compliance with the intervention protocol throughout the study duration.

Definitions

* Vitamin/Mineral Deficiency: For the purpose of this study, a deficiency is defined as a serum concentration below the lower limit of the standard laboratory reference range for that nutrient. Each participating laboratory will have established normal ranges for the measured vitamins and minerals; values below the 2.5th percentile of healthy individuals (the typical lower limit) will be considered deficient. For example, vitamin B_12 deficiency may be defined as B_12 < 200 pg/mL and vitamin D deficiency as 25-OHD < 20 ng/mL, based on commonly accepted thresholds, although the exact cut-off will depend on the assay reference range ￼. Participants will be considered to have a deficiency if any one or more of the tracked nutrients falls below the normal range at a given time point (excluding transient lab errors, which would be rechecked). Each distinct nutrient deficiency will also be recorded for analysis.
* Hypervitaminosis: Defined as a serum vitamin level above the upper limit of the normal reference range. For instance, vitamin B_6 above ~30 ng/mL or 25-OHD above ~100 ng/mL (depending on lab norms) would be flagged as potential hypervitaminosis. Any participant with a value above the normal range for a given vitamin at any time is noted as having hypervitaminosis (for that vitamin). The study intervention (Balance tablets) is formulated at standard recommended doses, so true hypervitaminosis is expected to be rare; however, tracking this ensures safety. If any levels are extremely high (e.g., >2 times upper limit), study clinicians will be notified to evaluate the participant for over-supplementation or other causes.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18-65 years.

  * BMI ≥ 30 kg/m² (obesity), or BMI ≥ 27 kg/m² with at least one obesity-related comorbidity (e.g., type 2 diabetes, hypertension).
  * Currently using a GLP-1 receptor agonist medication for weight management (e.g., semaglutide or liraglutide) and planning to continue it for the next year as part of their weight loss regimen.

Exclusion Criteria:

* • Any pre-existing condition that affects nutrient absorption or metabolism (e.g., malabsorptive gastrointestinal disorders such as celiac disease or inflammatory bowel disease, prior bariatric surgery).

  * Use of other weight loss medications (besides the GLP-1 RA) or use of high-dose vitamin/mineral supplements or other nutritional supplements that could influence vitamin/mineral status.
  * Pregnancy or lactation (women of childbearing potential will undergo a pregnancy test and must agree to use contraception during the study).
  * Known hypersensitivity or allergy to components of the Balance multivitamin formulation.
  * Significant chronic illnesses (e.g., end-stage renal disease, advanced liver disease) that in the investigator's judgment would interfere with participation or outcomes of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of vitamin and mineral deficiencies at 12 months, comparing the proportion of participants in each group who develop one or more deficiencies. | From enrollment to the end of treatment at 12 months
  Deficiency is defined for each nutrient as a serum concentration below the lower limit of the normal reference range (see Definitions below). The incidence of deficiencies will also be measured at interim time points (3, 6, and 9 months) to observe the trajectory over time, but the comparison at 12 months is the primary endpoint for efficacy.

SECONDARY OUTCOMES:
Serum nutrient levels | From enrollment to the end of treatment at 12 months
  Changes in specific vitamin and mineral concentrations from baseline at 3, 6, 9, and 12 months. This includes vitamins B_12, B_1 (thiamine), B_6 (pyridoxine), folic acid, 25-hydroxyvitamin D (25-OHD), and minerals such as iron stores (ferritin), calcium (albumin-corrected), magnesium, phosphate, zinc, as well as parathyroid hormone (PTH) and albumin (as a marker of nutritional status). For each of these analytes, the mean (or median) change over 12 months and the proportion of patients below normal range at each time point will be compared between groups.
Incidence of hypervitaminosis | From enrollment to the end of treatment at 12 months
  Number and proportion of participants in each group who develop hypervitaminosis (excess levels of any vitamin above the normal reference range) during the 12-month period. This will be assessed at the same blood sampling intervals. Particularly, fat-soluble vitamin levels (e.g., vitamins A, D, B_12) will be monitored for any values above the upper limit of normal.
Compliance with supplementation | From enrollment to the end of treatment at 12 months
  Adherence to the prescribed daily tablet regimen will be evaluated utilizing the 5-item Medication Adherence Report Scale (MARS-5), a validated instrument that identifies prevalent non-adherence patterns. Each of the five items will be rated on a 5-point Likert scale from 1 (indicating 'always') to 5 (indicating 'never'), yielding a cumulative score ranging from 5 to 25, where higher scores reflect improved adherence. At each designated follow-up interval (3, 6, 9, and 12 months), a bilingual study specialist will administer the MARS-5 questionnaire orally in the participant's preferred language, either Arabic or English, and meticulously document the responses. Comparative analyses of average adherence scores will be conducted between the Balance and placebo cohorts, and we will also assess the correlation between adherence levels and the occurrence of vitamin and mineral deficiencies.
Anthropometric outcome | From enrollment to the end of treatment at 12 months
  Changes in body weight and adiposity measure including BMI (weight and height will be combined to report BMI in kg/m^2) at 3, 6, 9, and 12 months. That outcome will indicate the degree of weight loss and will be tracked to ensure both groups have similar weight loss (since all are on GLP-1 therapy) and to explore if improved micronutrient status correlates with better weight outcomes or vice versa. (weight in kilograms, height in meters)
Anthropometric outcome | From enrollment to the end of treatment at 12 months
  Changes in body weight and adiposity measure including %EWL (weight in kilograms) at 3, 6, 9, and 12 months. %EWL is defined as the percentage of above-ideal body weight lost. That outcome will indicate the degree of weight loss and will be tracked to ensure both groups have similar weight loss (since all are on GLP-1 therapy) and to explore if improved micronutrient status correlates with better weight outcomes or vice versa.
Anthropometric outcome | From enrollment to the end of treatment at 12 months
  Changes in body weight and adiposity measure including %TWL (weight in kilograms) at 3, 6, 9, and 12 months. %TWL is the percentage of total body weight lost from baseline. These outcomes will indicate the degree of weight loss and will be tracked to ensure both groups have similar weight loss (since all are on GLP-1 therapy) and to explore if improved micronutrient status correlates with better weight outcomes or vice versa.

CONTACTS AND LOCATIONS:
Locations (1):
- Facility Name: The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Facility, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Whole study period
Access Criteria: Ask contact person